CLINICAL TRIAL: NCT00391534
Title: Safety and Efficacy of a Novel Modified Release Formulation of Oxcarbazepine (OXC MR) vs an Immediate Release Oxcarbazepine (OXC IR) Product in Patients With Partial Epilepsy
Brief Title: EXTENT: EXtended Tolerability and Efficacy of a Novel Formulation of Oxcarbazepine in a Trial in Partial Epilepsy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Desitin Arzneimittel GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Dr. Martina Wangemann, Desitin Arzneimittel GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXC-039/K; EudraCT No: 2006-003834-14
Record Dates: First submitted 2006-10-23; First posted 2006-10-24 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2009-01

CONDITIONS: Partial Epilepsy
Keywords: Epilepsy; oxcarbazepine
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxcarbazepine MR (Experimental): Patients who are pre-treated with a total daily dose of exactly 900 or exactly 1200 mg or exactly 1500 mg oxcarbazepine (as OXC IR) will increase dosage of OXC by 300 mg to a daily dose of 1200 mg / 1500 mg / 1800 mg OXC MR. Dosage will be titrated to a maximum tolerated total daily dose, maximally to 2700 mg in steps of 300 mg every 6th day.
  Interventions: Drug: modified release formulation of oxcarbazepine (OXC MR)
- Oxcarbazepine IR (Active Comparator): Patients who are pre-treated with a total daily dose of exactly 900 or exactly 1200 mg or exactly 1500 mg oxcarbazepine (as OXC IR) will increase dosage of OXC by 300 mg to a daily dose of 1200 mg / 1500 mg / 1800 mg OXC IR (divided in two daily doses). Dosage will be titrated to a maximum tolerated total daily dose, maximally to 2700 mg in steps of 300 mg every 6th day.
  Interventions: Drug: immediate release formulation of oxcarbazepine (OXC IR)

INTERVENTIONS:
Drug: modified release formulation of oxcarbazepine (OXC MR) — Patients who are pre-treated with a total daily dose of exactly 900 or exactly 1200 mg or exactly 1500 mg oxcarbazepine (as OXC IR) will increase dosage of OXC by 300 mg to a daily dose of 1200 mg / 1500 mg / 1800 mg OXC MR. Dosage will be titrated to a maximum tolerated total daily dose, maximally to 2700 mg in steps of 300 mg every 6th day.
  Arms: Oxcarbazepine MR
Drug: immediate release formulation of oxcarbazepine (OXC IR) — Patients who are pre-treated with a total daily dose of exactly 900 or exactly 1200 mg or exactly 1500 mg oxcarbazepine (as OXC IR) will increase dosage of OXC by 300 mg to a daily dose of 1200 mg / 1500 mg / 1800 mg OXC IR (divided in two daily doses). Dosage will be titrated to a maximum tolerated total daily dose, maximally to 2700 mg in steps of 300 mg every 6th day.
  Arms: Oxcarbazepine IR

SUMMARY:
This study is intended to investigate the safety and efficacy of a novel formulation of oxcarbazepine that is released more slowly than the current formulation. The study medication will be used as a treatment against partial epilepsy.

DETAILED DESCRIPTION:
This is a multi-centre, randomized, open-label, flexible-titration, controlled, parallel-group study to investigate the safety and efficacy of a novel modified release formulation of oxcarbazepine (OXC MR) compared to an immediate release oxcarbazepine (OXC IR) product in patients with partial epilepsy. Adult patients of both gender, aged at least 18 years with refractory partial epilepsy, with or without secondary generalisation receiving a stable background treatment with daily dosages of exactly 900 or 1200 or 1500 mg Oxcarbazepine will be enrolled. Concomitant medication consisting of maximal 2 additional AEDs (vagus nerve stimulator included) is allowed and must be kept stable throughout the study. Patients, who agree to participate, will first sign and date the informed consent and undergo an evaluation at screening visit to determine eligibility. Those patients who qualify will be enrolled in the study, assigned a patient ID, and will enter the 4-week baseline period. Each patient will receive a seizure diary to record the number of seizures during the baseline period. For Visit 1 the patient will return to the clinic and complete all baseline procedures. Patients who have met the entry criteria will be randomised. The two treatment groups consist of 50 patients each, one group to be treated with OXC MR b.i.d. and the other to be treated with OXC IR b.i.d. in a 1:1 randomization. Following assignment to one of both treatment groups the patient will enter the dose-titration phase. From Visit 1 (Study Day 1) a total daily dose of 1200 mg /1500 mg /1800 mg oxcarbazepine will be given to the randomised patients. From Day 6 the dosage will be titrated to a maximum total daily dose of 2700 mg in steps of 300 mg every 6th day. Patients who experienced intolerable adverse events could reduce their daily dose by 150 mg on the 2nd day of up-titration for the remainder of the treatment period. In case the reduced dosage will also not be tolerated, in a second step the dosage can be reduced by further 150 mg OXC. The maximal tolerated dose achieved on up-titration will be maintained up to the final visit (Study Day 26).

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients with minimal age of 18 years on the date of the first study visit.
* Stable treatment with Oxcarbazepine treatment (Timox® /Trileptal®), dosage: exactly 900 mg or exactly 1200 mg or exactly 1500 mg for at least 1 month prior to screening.
* >= 2 partial onset seizures with or without secondary generalisation refractory to existing AED therapy within the baseline period.
* Weight between >= 50 kg and < 100 kg.
* for females with child-bearing potential: negative pregnancy rest and highly effective form of birth control (females using hormonal contraceptives should use a different or additional means of birth control, e.g. IUD, abstinence, vasectomized partner, double barriere methods with or without oral contraceptives)
* Stable regimen of <= 2 concomitant AEDs (vagus nerve stimulator included) during the baseline period; lamotrigine dose may be adjusted at baseline.
* Ethnic origin: Caucasian.
* Subjects capable of complying with the study stipulations.
* Patients who have provided written informed consent to participate in this study.

Exclusion Criteria:

* Epilepsy secondary to progressive metabolic disease, malignant neoplasm, substance abuse, or active infection.
* Status epilepticus at any time during the baseline period.
* Lennox-Gastaut syndrome.
* Generalized epilepsy as primary diagnosis.
* Severe cardiac, pulmonary, haematological, hepatic, renal or neoplastic pathology.
* Acute medical conditions and/or conditions that could interfere with the absorption, metabolism or excretion of oxcarbazepine.
* History of clinically relevant psychiatric illness and/or drug abuse, drug addiction or alcoholism within the last 2 years.
* Treatment with psychotropic drugs, anticholinergic drugs, anti-parkinson medication, α1-antagonists, α2-antagonists, carbamazepine, topiramate, felbamate, vigabatrin. Stable treatment with selective serotonin-reuptake-inhibitor (SSRI) having been given for at least 4 weeks prior to screening as supportive treatment of partial epilepsy can be accepted.
* Intake of sodium lowering medication, e.g. diuretics and non-steroidal anti- inflammatory drugs. Occasional and short-term intake of non-steroidal anti- inflammatory drugs on demand (Ibuprofen, Paracetamol, ASS, Diclofenac and others) is allowed.
* Hypersensitivity towards oxcarbazepine or chemically related drugs.
* Low sodium serum levels (< 128 mmol/L). Sodium serum levels ≥ 126 and < 128 mmol/L can be accepted for inclusion, if these levels have been stable for at least 3 months.
* Symptomatic hyponatremia.
* Pregnancy or breast feeding.
* Participation in drug trials during 3 months preceding the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Maintenance dosage where dose up-titration has to be discontinued due to AEs | whenever criterion is met

SECONDARY OUTCOMES:
Number of seizures during the trial | Visit 1, Visit 2, Final Visit and each unscheduled visit
OXC and MHD plasma levels obtained from 6 patients per centre | Visit 1, Visit 2, Final Visit and each unscheduled visit
Adverse event profile Plus (AEP) questionnaire-score | at each patient contact
EpiTrack | Visit 1, Visit 2, Final Visit and each unscheduled visit
Vital Signs and ECG | Visit 1, Visit 2, Final Visit and each unscheduled visit
Laboratory parameters (hematology, serum chemistry, coagulation, urinalysis) | Visit 1, Visit 2, Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Christian E. Elger, Prof. MD, Principal Investigator — Klinik für Epileptologie, Universität Bonn, Bonn, Germany; Martina Wangemann, Dr., Study Director — Desitin Arzneimittel GmbH
Locations (6):
- Germany (6):
  - Bergisch Gladbach
  - Bonn
  - Erlangen
  - Freiburg im Breisgau
  - Göttingen
  - Kehl-Kork